CLINICAL TRIAL: NCT03569319
Title: The Development and Pilot Testing of Tailored Mediterranean Lifestyle Education to Encourage Behaviour Change in Participants With Subjective Cognitive Impairment
Brief Title: Tailored Mediterranean Lifestyle Education in Participants With Subjective Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Wellcome Trust (Other)
Responsible Party: Principal Investigator, Jayne Woodside, PhD, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18/NI/0077
Record Dates: First submitted 2018-06-03; First posted 2018-06-26 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Subjective Cognitive Impairment
Keywords: Mediterranean Diet; Lifestyle
MeSH Terms: interventions — BaseLine dental cement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: "THINK-MED" resource (baseline) (Experimental): The "THINK-MED" resource contains an information booklet, recipe books, menu plan cards, shopping list cards and goal setting cards. Participants will receive this resource on one occasion at baseline (n=10)
  Interventions: Behavioral: "THINK-MED" resource (baseline)
- Group 2: "THINK-MED" resource (staged) (Experimental): This group of participants will receive the "THINK-MED" resource at monthly intervals for 5 months accompanied by telephone feedback from the research dietitian (n=10)
  Interventions: Behavioral: "THINK-MED" resource (staged)
- Group 3: Control (Placebo Comparator): Participants will receive the "THINK-MED" resource after their final 6 month study visit (i.e. delayed intervention) (n=10)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: "THINK-MED" resource (baseline) — The "THINK-MED" resource contains an information booklet, recipe books, menu plan cards, shopping list cards and goal setting cards. Participants will receive this resource on one occasion at baseline.
  Arms: Group 1: "THINK-MED" resource (baseline)
Behavioral: "THINK-MED" resource (staged) — This group of participants will receive the "THINK-MED" resource at monthly intervals for 5 months accompanied by telephone feedback from the research dietitian
  Arms: Group 2: "THINK-MED" resource (staged)
Behavioral: Control — Participants will receive the "THINK-MED" resource after their final 6 month study visit (i.e. delayed intervention).
  Arms: Group 3: Control

SUMMARY:
It is estimated that 30% of Alzheimer's disease cases globally are associated with changeable risk factors, such as diet and physical activity. In particular, a Mediterranean diet (MD) has been associated with reduced risk of cognitive decline and improved brain function.

The investigators developed educational resources on the Mediterranean diet and lifestyle (THINK-MED) in accordance with the Medical Research Council guidance for developing and evaluating complex interventions, based on a systematic literature review and informed by qualitative work with patients with mild memory problems.The feedback gathered informed refinements and tailoring of the resource and overall MD intervention.

This study aims to evaluate feasibility of the "THINK-MED" Mediterranean lifestyle educational intervention to encourage dietary behaviour change among community-dwelling people with subjective cognitive impairment.

DETAILED DESCRIPTION:
This pilot RCT aims to evaluate the feasibility of a theory-based, tailored Mediterranean lifestyle education intervention (THINK-MED) to encourage behaviour change among participants who have subjective cognitive impairment.

This study will be a 6 month randomised controlled trial (RCT) with a total of 30 participants who will be randomised to 1 of 3 groups:

1. Group 1 will receive the "THINK-MED" Mediterranean Lifestyle Education for Memory resource on one occasion at baseline (n=10)
2. Group 2 will receive the "THINK-MED" Mediterranean Lifestyle Education for Memory resource at monthly intervals for 5 months, with an initial face-to-face visit from the research dietitian (month 1) and accompanied by telephone feedback (month 2-5) (n=10)
3. Group 3 is a control group. Participants in this group will receive the "THINK-MED" Mediterranean Lifestyle Education for Memory resource after completing the 6 month study (n=10)

ELIGIBILITY:
Inclusion Criteria:

* Have subjective cognitive impairment - Montreal Cognitive Assessment (MoCA) score ≥ 26/30
* Mediterranean diet score (MDS) ≤ 4 (Estruch et al. 2006)
* Willing to make changes to their diet

Exclusion Criteria:

* Diagnosis of dementia
* MoCA score of ≤ 25/30
* Individuals with a visual or English language impairment
* Psychiatric problems e.g. depression
* Significant medical comorbidity
* Body Mass Index (BMI) ≤ 19 and ≥ 40 kg/m2
* Excessive alcohol consumption
* Dietary restrictions/allergies that would substantially limit ability to complete study requirements
* Inability to provide informed consent
* History of, or comorbid condition which may alter performance on cognitive tests e.g. stroke, head injury, Parkinson's disease, learning disability

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Mediterranean Diet Score (MDS) at 6 months | Baseline, 6 months
  Mediterranean dietary intake will be measured by a validated questionnaire with a increase in score by greater than or equal to 3 points at 6 months indicating adoption (maximum score 14)

SECONDARY OUTCOMES:
Change in Physical Activity at 6 months | Baseline, 6 months
  Physical activity will be measured by the Recent Physical Activity Questionnaire (RPAQ)
Anthropometric measurements | Baseline, 6 months
  Weight and height measurements to calculate BMI
Muscle Strength | Baseline, 6 months
  Measured using a grip-strength dynamometer
Geriatric Depression Scale | Baseline, 6 months
  Depressive symptoms will be measured by the Geriatric Depression Scale Questionnaire, with a score greater than 5 indicating depressive symptoms
Functional Assessment (1) | Baseline, 6 months
  Measured by the instrumental activities of daily living questionnaire (IADL) by Lawton and Brody Measured by the instrumental activities of daily living scale (IADL) by Lawton and Brody (1969) questionnaire
Functional Assessment (2) | Baseline, 6 months
  Measured by the Bristol activities of daily living (Bucks et al. 1996) questionnaire
Cognitive Assessment | Baseline, 6 months
  A comprehensive cognitive assessment will be performed, including: global cognition, motor skills, executive function episodic/visual memory, and information processing and sustained attention using a validated neuropsychological test battery (Cantab Cognitive Battery, Cambridge Cognition Ltd.)
4 day food diary | Baseline, 6 months
  A food diary will be completed to assess compliance with a Mediterranean diet
Change in Lifestyle questionnaire | Baseline, 6 months
  A questionnaire to measure change in lifestyle behaviours
Dietary Quality of Life questionnaire | Baseline, 6 months
  A questionnaire to measure dietary quality of life
Mediterranean Diet Knowledge questionnaire | Baseline, 6 months
  A questionnaire to measure participants Mediterranean diet knowledge
Rand Short Form-36 HEALTH SURVEY | Baseline, 6 months
  A questionnaire to measure participants views and beliefs on health
Staging Algorithm Questionnaire | Baseline, 6 months
  A questionnaire to measure participants readiness to change their diet and lifestyle
Mediterranean Diet self-efficacy questionnaire | Baseline, 6 months
  A questionnaire to measure participants self-efficacy
Barriers to consuming a Mediterranean Diet questionnaire | Baseline, 6 months
  Dietary behaviour change questionnaire to measure adherence to a Mediterranean diet
Blood Sample | Baseline, 6 months
  A blood sample will be taken from participants to be stored for analysis of biomarkers of MD adherence and biomarkers of neurodegenerative disease risk.

OTHER OUTCOMES:
Process Evaluation (1) - telephone contact evaluation | Up to 3 months post intervention
  Determination individual participation and engagement with the intervention by reviewing telephone contact log record and telephone checklist evaluation
Process Evaluation (2) - study records | Up to 3 months post intervention
  A review of study records- including attrition rates, reason for dropout
Process Evaluation (3) - structured interviews | Up to 3 months post intervention
  Post intervention structured interviews for participant evaluation of the intervention programme and dietary educational materials

CONTACTS AND LOCATIONS:
Overall Officials: Jayne Woodside, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Queen's University, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] McGrattan AM, McEvoy CT, Vijayakumar A, Moore SE, Neville CE, McGuinness B, McKinley MC, Woodside JV. A mixed methods pilot randomised controlled trial to develop and evaluate the feasibility of a Mediterranean diet and lifestyle education intervention 'THINK-MED' among people with cognitive impairment. Pilot Feasibility Stud. 2021 Jan 4;7(1):3. doi: 10.1186/s40814-020-00738-3. PMID 33390187